CLINICAL TRIAL: NCT02181738
Title: Non-Comparative, Multi-Cohort, Single Arm, Open-Label, Phase 2 Study of Nivolumab (BMS-936558) in Classical Hodgkin Lymphoma (cHL) Subjects
Brief Title: Study of Nivolumab in Patients With Classical Hodgkin's Lymphoma (Registrational)
Acronym: CheckMate 205
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-205; 2014-001509-42 (EudraCT Number)
Record Dates: First submitted 2014-07-01; First posted 2014-07-04 (Estimated); Results first posted 2018-12-11 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Hodgkin Disease
MeSH Terms: conditions — Hodgkin Disease | interventions — Nivolumab; Doxorubicin; Vinblastine; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nivolumab (Cohort A, B, C and D) (Experimental): Cohort (A, B, C): Nivolumab: Specified dose on specified days
  Cohort (D): Nivolumab: Specified dose on specified days + Doxorubicin: Specified dose on specified days + Vinblastine: Specified dose on specified days + Dacarbazine: Specified dose on specified days
  Interventions: Drug: Nivolumab; Drug: Doxorubicin; Drug: Vinblastine; Drug: Dacarbazine

INTERVENTIONS:
Drug: Nivolumab — Specified dose on specified days
  Other Names: BMS-936558
Drug: Doxorubicin — Specified dose on specified days
Drug: Vinblastine — Specified dose on specified days
Drug: Dacarbazine — Specified dose on specified days

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Nivolumab in previously treated (cohorts, A, B & C) or newly diagnosed (cohort D) classical Hodgkin Lymphoma participants.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Must have received prior high-dose conditioning chemotherapy followed by autologous stem cell transplant (ASCT) as a part of salvage therapy for cHL (cohort A, B & C - enrollment closed)
* Participants may be Brentuximab vedotin- naïve, or may have had prior Brentuximab vedotin treatment (cohort A, B & C - enrollment closed)
* Newly diagnosed and previously untreated classical Hodgkin Lymphoma (cohort D)

Exclusion Criteria:

* Known central nervous system lymphoma
* Participants with nodular lymphocyte-predominant Hodgkin Lymphoma
* Prior allogeneic stem cell transplantation (SCT)
* Chest radiation ≤ 24 weeks prior to first dose
* Carmustine ≥ 600 mg/m² received as part of the pre-transplant conditioning regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2014-08-12 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2022-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (38):
- United States (14):
  - Local Institution - 0030, Los Angeles, California
  - Local Institution - 0009, Los Angeles, California
  - Local Institution - 0001, Atlanta, Georgia
  - Local Institution - 0002, Boston, Massachusetts
  - Local Institution - 0025, Boston, Massachusetts
  - Local Institution - 0041, Boston, Massachusetts
  - Local Institution - 0008, Detroit, Michigan
  - Local Institution - 0003, Rochester, Minnesota
  - Local Institution - 0047, Hackensack, New Jersey
  - Local Institution - 0040, Basking Ridge, New York
  - Local Institution - 0005, New York, New York
  - Local Institution - 0006, Allentown, Pennsylvania
  - Local Institution - 0004, Nashville, Tennessee
  - Local Institution - 0007, Houston, Texas
- Austria (2):
  - Local Institution - 0032, Innsbruck
  - Local Institution - 0031, Vienna
- Belgium (2):
  - Local Institution - 0014, B-leuven
  - Local Institution - 0015, Ghent
- Canada (2):
  - Local Institution - 0046, Vancouver, British Columbia
  - Local Institution - 0042, Toronto, Ontario
- Local Institution - 0044, Prague, Czechia
- Germany (4):
  - Local Institution - 0037, Berlin
  - Local Institution - 0033, Cologne
  - Local Institution - 0036, Hamburg
  - Local Institution - 0034, Ulm
- Italy (3):
  - Local Institution - 0019, Bologna
  - Local Institution - 0020, Napoli
  - Local Institution - 0035, Rozzano (milano)
- Netherlands (3):
  - Local Institution - 0016, Amsterdam
  - Local Institution - 0038, Groningen
  - Local Institution - 0017, Utrecht
- Spain (3):
  - Local Institution - 0022, Hospitalet Llobregat- Barcelona
  - Local Institution - 0027, Majadahonda - Madrid
  - Local Institution - 0023, Marbella
- United Kingdom (4):
  - Local Institution - 0043, Swansea, Carmarthenshire
  - Local Institution - 0012, Withington, Manchester
  - Local Institution - 0026, Oxford, Oxfordshire
  - Local Institution - 0013, Sutton

REFERENCES:
- [Derived] Cader FZ, Hu X, Goh WL, Wienand K, Ouyang J, Mandato E, Redd R, Lawton LN, Chen PH, Weirather JL, Schackmann RCJ, Li B, Ma W, Armand P, Rodig SJ, Neuberg D, Liu XS, Shipp MA. A peripheral immune signature of responsiveness to PD-1 blockade in patients with classical Hodgkin lymphoma. Nat Med. 2020 Sep;26(9):1468-1479. doi: 10.1038/s41591-020-1006-1. Epub 2020 Aug 10. PMID 32778827
- [Derived] Ramchandren R, Domingo-Domenech E, Rueda A, Trneny M, Feldman TA, Lee HJ, Provencio M, Sillaber C, Cohen JB, Savage KJ, Willenbacher W, Ligon AH, Ouyang J, Redd R, Rodig SJ, Shipp MA, Sacchi M, Sumbul A, Armand P, Ansell SM. Nivolumab for Newly Diagnosed Advanced-Stage Classic Hodgkin Lymphoma: Safety and Efficacy in the Phase II CheckMate 205 Study. J Clin Oncol. 2019 Aug 10;37(23):1997-2007. doi: 10.1200/JCO.19.00315. Epub 2019 May 21. PMID 31112476
- [Derived] Armand P, Engert A, Younes A, Fanale M, Santoro A, Zinzani PL, Timmerman JM, Collins GP, Ramchandren R, Cohen JB, De Boer JP, Kuruvilla J, Savage KJ, Trneny M, Shipp MA, Kato K, Sumbul A, Farsaci B, Ansell SM. Nivolumab for Relapsed/Refractory Classic Hodgkin Lymphoma After Failure of Autologous Hematopoietic Cell Transplantation: Extended Follow-Up of the Multicohort Single-Arm Phase II CheckMate 205 Trial. J Clin Oncol. 2018 May 10;36(14):1428-1439. doi: 10.1200/JCO.2017.76.0793. Epub 2018 Mar 27. PMID 29584546
- [Derived] Roemer MGM, Redd RA, Cader FZ, Pak CJ, Abdelrahman S, Ouyang J, Sasse S, Younes A, Fanale M, Santoro A, Zinzani PL, Timmerman J, Collins GP, Ramchandren R, Cohen JB, De Boer JP, Kuruvilla J, Savage KJ, Trneny M, Ansell S, Kato K, Farsaci B, Sumbul A, Armand P, Neuberg DS, Pinkus GS, Ligon AH, Rodig SJ, Shipp MA. Major Histocompatibility Complex Class II and Programmed Death Ligand 1 Expression Predict Outcome After Programmed Death 1 Blockade in Classic Hodgkin Lymphoma. J Clin Oncol. 2018 Apr 1;36(10):942-950. doi: 10.1200/JCO.2017.77.3994. Epub 2018 Feb 2. PMID 29394125
- [Derived] Hude I, Sasse S, Brockelmann PJ, von Tresckow B, Momotow J, Engert A, Borchmann S. Leucocyte and eosinophil counts predict progression-free survival in relapsed or refractory classical Hodgkin Lymphoma patients treated with PD1 inhibition. Br J Haematol. 2018 Jun;181(6):837-840. doi: 10.1111/bjh.14705. Epub 2017 Apr 25. No abstract available. PMID 28439879
- [Derived] Younes A, Santoro A, Shipp M, Zinzani PL, Timmerman JM, Ansell S, Armand P, Fanale M, Ratanatharathorn V, Kuruvilla J, Cohen JB, Collins G, Savage KJ, Trneny M, Kato K, Farsaci B, Parker SM, Rodig S, Roemer MG, Ligon AH, Engert A. Nivolumab for classical Hodgkin's lymphoma after failure of both autologous stem-cell transplantation and brentuximab vedotin: a multicentre, multicohort, single-arm phase 2 trial. Lancet Oncol. 2016 Sep;17(9):1283-94. doi: 10.1016/S1470-2045(16)30167-X. Epub 2016 Jul 20. PMID 27451390
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 243 participants were treated at 34 sites in 10 countries for cohorts A, B, and C. Cohort D enrolled separately. 51 participants were treated in cohort D for a total of 294 participants treated all together.
Groups:
- Cohort A: Post-Transplant, Never Taken Brentuximab Vedotin; Cohort B: Post Transplant, Brentuximab Vedotin Taken Post-Autologous Stem Cell Transplant; Cohort C: Post Transplant, Brentuximab Vedotin Taken Pre-and/or Post-Autologous Stem Cell Transplant: Nivolumab was administered at 3 mg/kg IV over 60 minutes on the first day of each 2-week cycle. Upon the implementation of revised protocol version 04c (dated 22-Aug-2019), participants were switched from a body weight-based dose of 3 mg/kg every 2 weeks to a flat dose of 480 mg every 4 weeks or a flat dose of 240 mg every 2 weeks. Nivolumab treatment was continued until unacceptable toxicity or disease progression.
- Cohort D: Newly Diagnosed, Previously Untreated Advanced Stage cHL (Stage IIB, III and IV): Four doses of nivolumab flat dose 240 mg IV were administered every 2 weeks (monotherapy phase), followed by 12 doses of the combination of AVD (adriamycin/ doxorubicin 25 mg/m2, vinblastine 6 mg/m2, dacarbazine 375 mg/m2) chemotherapy and nivolumab flat dose 240 mg IV for 6 cycles (combination phase).
Period: Overall Study
Arm/Group | Cohort A: Post-Transplant, Never Taken Brentuximab Vedotin | Cohort B: Post Transplant, Brentuximab Vedotin Taken Post-Autologous Stem Cell Transplant | Cohort C: Post Transplant, Brentuximab Vedotin Taken Pre-and/or Post-Autologous Stem Cell Transplant | Cohort D: Newly Diagnosed, Previously Untreated Advanced Stage cHL (Stage IIB, III and IV)
Started | 63 | 80 | 100 | 51
N-AVD Combination Therapy Phase (Received N-AVD) | 0 | 0 | 0 | 49
N-AVD Combination Therapy Phase (Received only AVD) | 0 | 0 | 0 | 1
Completed (Completed = completed treatment as per protocol) | 0 | 0 | 13 | 45
Not Completed | 63 | 80 | 87 | 6
Not completed — Participant Withdrew Consent | 2 | 1 | 1 | 1
Not completed — Lost to Follow-up | 1 | 2 | 1 | 1
Not completed — Participant no Longer Meets Study Criteria | 0 | 0 | 0 | 1
Not completed — Poor/Non-Compliance | 1 | 0 | 2 | 1
Not completed — Disease Progression | 28 | 35 | 40 | 0
Not completed — Participant Request to Discontinue Study Treatment | 5 | 12 | 5 | 1
Not completed — Study Drug Toxicity | 6 | 11 | 8 | 1
Not completed — Other Reasons | 14 | 16 | 28 | 0
Not completed — Maximum Clinical Benefit | 3 | 0 | 1 | 0
Not completed — Adverse Event Unrelated to Study Drug | 3 | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Post-Transplant, Never Taken Brentuximab Vedotin | Cohort B: Post Transplant, Brentuximab Vedotin Taken Post-Autologous Stem Cell Transplant | Cohort C: Post Transplant, Brentuximab Vedotin Taken Pre-and/or Post-Autologous Stem Cell Transplant | Cohort D: Newly Diagnosed, Previously Untreated Advanced Stage cHL (Stage IIB, III and IV) | Total
Number analyzed (Participants) | 63 | 80 | 100 | 51 | 294
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: All treated participants
  Years | 36.3 (12.54) | 38.7 (13.00) | 36.1 (12.41) | 39.0 (16.88) | 37.4 (13.47)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All treated participants
  Participants
    Female | 29 | 29 | 44 | 19 | 121
    Male | 34 | 51 | 56 | 32 | 173
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: All treated participants
  Participants
    Hispanic or Latino | 3 | 1 | 1 | 0 | 5
    Not Hispanic or Latino | 30 | 63 | 56 | 40 | 189
    Unknown or Not Reported | 30 | 16 | 43 | 11 | 100
Race/Ethnicity, Customized [Number; unit: Participants] — Population: All treated particpants
  Participants
    White | 54 | 71 | 86 | 45 | 256
    Black or African | 2 | 4 | 6 | 2 | 14
    Asian | 3 | 1 | 5 | 2 | 11
    American Indian or Alaska Native | 0 | 0 | 2 | 0 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Other | 4 | 4 | 1 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Based on IRRC Assessments in Cohorts A, B, and C
Description: ORR is the percent of participants achieving either a complete remission (CR) or partial remission (PR) according to the 2007 IWG criteria. Analyses of efficacy endpoints were performed separately for each cohort, according to IWG 2007. For cohort A and B, if the bone marrow was involved by lymphoma before treatment, the infiltrate must have cleared on repeat bone marrow biopsy. For cohort C, no evidence of FDG-avid disease in bone marrow was required in all participants in lieu of bone marrow aspirate/ biopsy.
  CR is the percent of participants with a best overall response (BOR) of CR (disappearance of all evidence of disease) according to the 2007 IWG criteria, based on IRRC assessment.
  PR is the percent of participants with a best overall response (BOR) of PR (regression of measurable disease and no new sites) according to the 2007 IWG criteria, based on IRRC assessment.
  Confidence interval based on Clopper-Pearson method.
Time Frame: From first dose to the date of initial objectively documented progression or the date of subsequent therapy, whichever occurred first (up to approximately 28 months)
Population: All treated Cohort A, B and C participants
Measure: Number (95% Confidence Interval); unit: Percentage of Particpants
Arm/Group | Cohort A: Post-Transplant, Never Taken Brentuximab Vedotin | Cohort B: Post Transplant, Brentuximab Vedotin Taken Post-Autologous Stem Cell Transplant | Cohort C: Post Transplant, Brentuximab Vedotin Taken Pre-and/or Post-Autologous Stem Cell Transplant
Number analyzed (Participants) | 63 | 80 | 100
Percentage of Particpants | 65.1 [52.0 to 76.7] | 67.5 [56.1 to 77.6] | 73.0 [63.2 to 81.4]

2. Primary Outcome: Number of Participants Who Experienced at Least One Treatment Related Grade 3-5 AE in Cohort D
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation subject administered study drug and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug.
Time Frame: From first dose of the considered therapy phase to 30 days after last dose of study therapy phase (or up to first dose of combination if any when considering the monotherapy period) (an average of 8 months and a maximum of 11 months)
Population: All Cohort D participants treated in the monotherapy and combination therapy phases.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D: Newly Diagnosed, Previously Untreated Advanced Stage cHL (Stage IIB, III and IV)
Number analyzed (Participants) | 51
Participants
  Monotherapy | 0
  Combination Therapy (receiving AVD or NAVD): number analyzed (Participants) | 50
  Combination Therapy (receiving AVD or NAVD) | 30

3. Secondary Outcome: Duration of Objective Response Based on IRRC Assessments in Cohorts A, B, and C
Description: DOR is the time from first response (complete remission (CR) or partial remission (PR)) to the date of initial objectively documented progression as determined using the 2007 IWG criteria or death due to any cause, whichever occurred first. For participants who neither progressed nor died, the DOR was censored on the date of their last tumor assessment. Participants who started subsequent therapy without a prior reported progression were censored at the last tumor assessments prior to initiation of the subsequent anticancer therapy.
  CR is the percent of participants with a best overall response (BOR) of CR (disappearance of all evidence of disease) according to the 2007 IWG criteria, based on IRRC assessment.
  PR is the percent of participants with a best overall response (BOR) of PR (regression of measurable disease and no new sites) according to the 2007 IWG criteria, based on IRRC assessment.
  Computed using Kaplan-Meier method.
Time Frame: From first dose to the date of initial objectively documented progression or the date of subsequent therapy, or death whichever occurred first (up to approximately 100 months).
Population: All treated Cohort A, B and C participants with objective response of CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Post-Transplant, Never Taken Brentuximab Vedotin | Cohort B: Post Transplant, Brentuximab Vedotin Taken Post-Autologous Stem Cell Transplant | Cohort C: Post Transplant, Brentuximab Vedotin Taken Pre-and/or Post-Autologous Stem Cell Transplant
Number analyzed (Participants) | 41 | 57 | 75
Months | 26.18 [15.21 to NA] — The upper 95% confidence interval was not reached due to Insufficient number of participants with events to reach the threshold according to Kaplan-Meier methodology. | 16.59 [9.26 to 25.72] | 18.17 [11.63 to 30.85]

4. Secondary Outcome: Complete Remission (CR) Rate Based on IRRC Assessments in Cohorts A, B, and C
Description: The CR rate was defined as the percent of participants with a BOR of CR (disappearance of all evidence of disease) according to the 2007 IWG criteria, based on IRRC assessment.
  Confidence interval based on Clopper-Pearson method.
Time Frame: as for outcome 3
Population: All treated Cohort A, B and C participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Post-Transplant, Never Taken Brentuximab Vedotin | Cohort B: Post Transplant, Brentuximab Vedotin Taken Post-Autologous Stem Cell Transplant | Cohort C: Post Transplant, Brentuximab Vedotin Taken Pre-and/or Post-Autologous Stem Cell Transplant
Number analyzed (Participants) | 63 | 80 | 100
Percentage of Participants | 31.7 [20.6 to 44.7] | 13.8 [7.1 to 23.3] | 21 [13.5 to 30.3]

5. Secondary Outcome: Duration of Complete Remission (CR) Based on IRRC Assessments for Cohorts A, B, and C
Description: The duration of CR was only evaluated in participants with BOR of CR and was defined as the time from first documentation of CR (the date of first negative FDG-PET scan or the date of first documentation of no disease involvement in the bone marrow (if required), whichever occurred later) to the date of initial objectively documented progression (Any new lesion or increase by >=50% of previously involved sites from nadir) as determined using the 2007 IWG criteria or death due to any cause, whichever occurred first. Censoring was applied as per DOR definition.
  Computed using Kaplan-Meier method.
Time Frame: as for outcome 3
Population: All treated Cohort A, B and C participants who had a BOR of CR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Post-Transplant, Never Taken Brentuximab Vedotin | Cohort B: Post Transplant, Brentuximab Vedotin Taken Post-Autologous Stem Cell Transplant | Cohort C: Post Transplant, Brentuximab Vedotin Taken Pre-and/or Post-Autologous Stem Cell Transplant
Number analyzed (Participants) | 20 | 11 | 21
Months | 43.47 [18.00 to NA] — The upper 95% confidence interval was not reached due to Insufficient number of participants with events to reach the threshold according to Kaplan-Meier methodology. | 30.32 [2.4 to NA] — The upper 95% confidence interval was not reached due to Insufficient number of participants with events to reach the threshold according to Kaplan-Meier methodology. | 26.41 [7.13 to NA] — The upper 95% confidence interval was not reached due to Insufficient number of participants with events to reach the threshold according to Kaplan-Meier methodology.

6. Secondary Outcome: Partial Remission (PR) Rate Based on IRRC Assessments in Cohorts A, B, and C
Description: The PR rate was defined as the percent of participants with a BOR of PR (regression of measurable disease and no new sites) according to the 2007 IWG criteria, based on IRRC assessment.
  Confidence interval based on Clopper-Pearson method.
Time Frame: as for outcome 3
Population: All treated Cohort A, B and C participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Post-Transplant, Never Taken Brentuximab Vedotin | Cohort B: Post Transplant, Brentuximab Vedotin Taken Post-Autologous Stem Cell Transplant | Cohort C: Post Transplant, Brentuximab Vedotin Taken Pre-and/or Post-Autologous Stem Cell Transplant
Number analyzed (Participants) | 63 | 80 | 100
Percentage of Participants | 33.3 [22.0 to 46.3] | 57.5 [45.9 to 68.5] | 54.0 [43.7 to 64.0]

7. Secondary Outcome: Duration of PR Based on IRRC Assessments in Cohorts A, B, and C
Description: The duration of PR was only evaluated in participants with BOR of PR and was defined as the time from first documentation of PR (regression of measurable disease and no new sites) to the date of initial objectively documented progression (any new lesion or increase by >=50% of previously involved sites from nadir) as determined using the 2007 IWG criteria or death due to any cause, whichever occurred first. Censoring was applied as per DOR definition.
  Computed using Kaplan-Meier method.
Time Frame: as for outcome 3
Population: All treated Cohort A, B and C participants who had a BOR of PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Post-Transplant, Never Taken Brentuximab Vedotin | Cohort B: Post Transplant, Brentuximab Vedotin Taken Post-Autologous Stem Cell Transplant | Cohort C: Post Transplant, Brentuximab Vedotin Taken Pre-and/or Post-Autologous Stem Cell Transplant
Number analyzed (Participants) | 21 | 46 | 54
Months | 12.78 [4.17 to 27.17] | 10.58 [7.46 to 25.26] | 14.65 [9.36 to 30.36]

8. Secondary Outcome: Objective Response Rates (ORR) Based on Investigator Assessments for Cohorts A, B, and C
Description: as for outcome 1
Time Frame: as for outcome 3
Population: All treated Cohort A, B and C participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Post-Transplant, Never Taken Brentuximab Vedotin | Cohort B: Post Transplant, Brentuximab Vedotin Taken Post-Autologous Stem Cell Transplant | Cohort C: Post Transplant, Brentuximab Vedotin Taken Pre-and/or Post-Autologous Stem Cell Transplant
Number analyzed (Participants) | 63 | 80 | 100
Percentage of Participants | 69.8 [57.0 to 80.8] | 73.8 [62.7 to 83.0] | 70.0 [60.0 to 78.8]

9. Secondary Outcome: Duration of Objective Response (DOR) Based on Investigator Assessments in Cohorts A, B, and C
Description: as for outcome 3
Time Frame: as for outcome 3
Population: All treated Cohort A, B and C participants who had a BOR of CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Post-Transplant, Never Taken Brentuximab Vedotin | Cohort B: Post Transplant, Brentuximab Vedotin Taken Post-Autologous Stem Cell Transplant | Cohort C: Post Transplant, Brentuximab Vedotin Taken Pre-and/or Post-Autologous Stem Cell Transplant
Number analyzed (Participants) | 44 | 59 | 70
Months | 39.10 [16.59 to 78.29] | 25.26 [10.09 to 41.72] | 28.85 [12.02 to 34.53]

10. Secondary Outcome: Treatment Discontinuation Rate in Cohort D
Description: Treatment discontinuation rate (TDR) is the number of treated participants who received <4 doses of monotherapy or <12 doses of their assigned combination regimen. A participant is considered as having received an AVD/NAVD dose as soon as they received at least one drug of AVD/NAVD for the considered dose. Participants must have received at least one dose of Nivolumab during the combination therapy phase to be included in participants treated with NAVD. If a participant subsequently met Criteria to Resume Nivolumab Dosing, the combination of nivolumab and AVD could be used. Participants who underwent treatment beyond progression during the Monotherapy phase could use the combination of nivolumab and AVD if all 4 doses of nivolumab monotherapy are completed.
  Discontinuation can be due to any reason including, but not limited to, drug-related toxicity, diseases progression, or death.
Time Frame: From first dose up until the date of treatment discontinuation (up to approximately 100 months).
Population: All Cohort D participants treated in the monotherapy and combination therapy phases.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D: Newly Diagnosed, Previously Untreated Advanced Stage cHL (Stage IIB, III and IV)
Number analyzed (Participants) | 51
Participants
  Monotherapy | 2
  Combination Therapy (receiving AVD or NAVD): number analyzed (Participants) | 50
  Combination Therapy (receiving AVD or NAVD) | 5
  Combination Therapy (NAVD receivers only): number analyzed (Participants) | 49
  Combination Therapy (NAVD receivers only) | 5
  Overall Therapy | 6

11. Secondary Outcome: Number of Participants Who Died in Cohort D
Description: Number of participants who died in Cohort D within 100 days after last dose of study therapy.
Time Frame: From first dose of the considered therapy phase to 100 days after last dose of study therapy phase (or up to first dose of combination if any when considering the monotherapy period) (an average of 10 months up to a maximum of 13 months)
Population: All Cohort D participants treated in the monotherapy and combination therapy phases.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D: Newly Diagnosed, Previously Untreated Advanced Stage cHL (Stage IIB, III and IV)
Number analyzed (Participants) | 51
Participants
  Monotherapy | 0
  Combination Therapy (receiving AVD or NAVD): number analyzed (Participants) | 50
  Combination Therapy (receiving AVD or NAVD) | 1

12. Secondary Outcome: Number of Participants With Adverse Events (AEs) in Cohort D
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study drug and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. Toxicities were graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: as for outcome 2
Population: All treated participants in Cohort D
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D: Newly Diagnosed, Previously Untreated Advanced Stage cHL (Stage IIB, III and IV)
Number analyzed (Participants) | 51
Participants
  Monotherapy | 48
  Combination Therapy (receiving AVD or NAVD): number analyzed (Participants) | 50
  Combination Therapy (receiving AVD or NAVD) | 49

13. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) in Cohort D
Description: A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose results in death, is life-threatening (defined as an event in which the participant was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe), requires inpatient hospitalization or causes prolongation of existing hospitalization. Toxicities were graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: as for outcome 2
Population: All treated participants in Cohort D
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D: Newly Diagnosed, Previously Untreated Advanced Stage cHL (Stage IIB, III and IV)
Number analyzed (Participants) | 51
Participants
  Monotherapy | 2
  Combination Therapy (receiving AVD or NAVD): number analyzed (Participants) | 50
  Combination Therapy (receiving AVD or NAVD) | 10

14. Secondary Outcome: Number of Participants With AEs Leading to Discontinuation in Cohort D
Description: as for outcome 12
Time Frame: as for outcome 2
Population: All treated participants in Cohort D
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D: Newly Diagnosed, Previously Untreated Advanced Stage cHL (Stage IIB, III and IV)
Number analyzed (Participants) | 51
Participants
  Monotherapy | 1
  Combination Therapy (receiving AVD or NAVD): number analyzed (Participants) | 50
  Combination Therapy (receiving AVD or NAVD) | 3

15. Secondary Outcome: Number of Participants With AEs Leading to Dose Delay in Cohort D
Description: as for outcome 12
Time Frame: as for outcome 2
Population: All treated participants in Cohort D
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D: Newly Diagnosed, Previously Untreated Advanced Stage cHL (Stage IIB, III and IV)
Number analyzed (Participants) | 51
Participants
  Monotherapy | 3
  Combination Therapy (receiving AVD or NAVD): number analyzed (Participants) | 50
  Combination Therapy (receiving AVD or NAVD) | 29

16. Secondary Outcome: Number of Participants With Select AEs in Cohort D
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study drug and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (such as an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not considered related to the study drug. Toxicities were graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Select AEs have been categorized into seven areas: pulmonary toxicity, gastrointestinal toxicity, hepatotoxicity, endocrinopathy, skin toxicity, neurological toxicity and renal toxicity. Select AEs, in particular pneumonitis, are considered clinically meaningful as they require greater vigilance and for early recognition and prompt intervention.
Time Frame: as for outcome 2
Population: All treated participants in Cohort D
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D: Newly Diagnosed, Previously Untreated Advanced Stage cHL (Stage IIB, III and IV)
Number analyzed (Participants) | 51
Participants
  Gastrointestinal Monotherapy | 6
  Gastrointestinal Combination Therapy | 13
  Hepatic Monotherapy | 2
  Hepatic Combination Therapy | 3
  Pulmonary Monotherapy | 0
  Pulmonary Combination Therapy | 3
  Renal Monotherapy | 1
  Renal Combination Therapy | 0
  Skin Monotherapy | 17
  Skin Combination Therapy | 9
  Hypersensitivity/Infusion Reactions Monotherapy | 16
  Hypersensitivity/Infusion Reactions Combination | 4

17. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Specific Thyroid Tests in Cohort D Monotherapy Phase
Description: The number of participants with laboratory abnormalities in specific thyroid tests based on SI conventional units. TSH = Thyroid Stimulating Hormone LLN = Lower Limit of Normal ULN = Upper Limit of Normal
Time Frame: From first dose of monotherapy to 30 days after last dose of monotherapy phase (up to approximately 3 months)
Population: All participants treated in the Cohort D monotherapy phase who had at least one on-treatment TSH measurement during the monotherapy phase
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D: Newly Diagnosed, Previously Untreated Advanced Stage cHL (Stage IIB, III and IV)
Number analyzed (Participants) | 42
Participants
  TSH > ULN | 1
  TSH > ULN WITH TSH <= ULN AT BASELINE | 1
  TSH >ULN WITH ATLEAST ONE FT3/FT4 TEST VALUE <LLN | 0
  TSH >ULN WITH ALL OTHER FT3/FT4 TEST VALUES >= LLN | 0
  TSH > ULN WITH FT3/FT4 TEST MISSING | 1
  TSH < LLN | 5
  TSH <LLN WITH TSH >= LLN AT BASELINE | 5
  TSH <LLN WITH ATLEAST ONE FT3/FT4 TEST VALUE > ULN | 1
  TSH <LLN WITH ALL OTHER FT3/FT4 TEST VALUES <= ULN | 0
  TSH < LLN WITH FT3/FT4 TEST MISSING | 4

18. Secondary Outcome: Number of Participants Laboratory Abnormalities in Specific Thyroid Tests in Cohort D Combination Therapy Phase
Description: as for outcome 17
Time Frame: From first dose of the combination therapy to 30 days after last dose of combination therapy (an average of 8 months and a maximum of 11 months)
Population: All participants treated in the Cohort D combination therapy phase who had at least one on-treatment AST, ALT and/or bilirubin test measurement during the combination therapy phase
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D: Newly Diagnosed, Previously Untreated Advanced Stage cHL (Stage IIB, III and IV)
Number analyzed (Participants) | 48
Participants
  TSH > ULN | 12
  TSH > ULN WITH TSH <= ULN AT BASELINE | 8
  TSH >ULN WITH ATLEAST ONE FT3/FT4 TEST VALUE <LLN | 3
  TSH >ULN WITH ALL OTHER FT3/FT4 TEST VALUES >= LLN | 1
  TSH > ULN WITH FT3/FT4 TEST MISSING | 8
  TSH < LLN | 5
  TSH <LLN WITH TSH >= LLN AT BASELINE | 5
  TSH <LLN WITH ATLEAST ONE FT3/FT4 TEST VALUE > ULN | 1
  TSH <LLN WITH ALL OTHER FT3/FT4 TEST VALUES <= ULN | 0
  TSH < LLN WITH FT3/FT4 TEST MISSING | 4

19. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Specific Liver Tests in Cohort D Monotherapy Phase
Description: The number of participants with laboratory abnormalities in specific liver tests based on SI conventional units. ALT = Alanine Aminotransferase, AST = Aspartate Aminotransferase, ULN = Upper Limit of Normal.
Time Frame: From first dose of monotherapy to 30 days after last dose of monotherapy phase (up to approximately 3 months)
Population: All participants treated in the Cohort D monotherapy phase
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D: Newly Diagnosed, Previously Untreated Advanced Stage cHL (Stage IIB, III and IV)
Number analyzed (Participants) | 51
Participants
  ALT OR AST > 3XULN | 2
  ALT OR AST> 5XULN | 1
  ALT OR AST> 10XULN | 0
  ALT OR AST > 20XULN | 0
  TOTAL BILIRUBIN > 2XULN | 0
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>2XULN IN 1 DAY | 0
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>2XULN IN 30 DAYS | 0

20. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Specific Liver Tests in Cohort D Combination Therapy Phase
Description: as for outcome 19
Time Frame: as for outcome 18
Population: All participants treated in the Cohort D combination therapy phase with at least one on-treatment laboratory measurement
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort D: Newly Diagnosed, Previously Untreated Advanced Stage cHL (Stage IIB, III and IV)
Number analyzed (Participants) | 49
Participants
  ALT OR AST > 3XULN | 4
  ALT OR AST> 5XULN | 1
  ALT OR AST> 10XULN | 1
  ALT OR AST > 20XULN | 0
  TOTAL BILIRUBIN > 2XULN | 0
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>2XULN IN 1 DAY | 0
  ALT/AST ELEV>3XULN;TOTAL BILIRUBIN>2XULN IN 30 DAYS | 0

21. Secondary Outcome: Complete Response (CR) Rate at Planned End of Therapy Based on IRRC Assessments in Cohort D
Description: CR rate is the percent of participants who show CR (disappearance of all evidence of disease) according to the 2007 IWG criteria at the planned end of study therapy radiographic tumor assessment.
  Confidence interval based on the Klopper and Pearson method.
Time Frame: as for outcome 3
Population: All Cohort D participants treated in the monotherapy and combination therapy phases.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Cohort D: Newly Diagnosed, Previously Untreated Advanced Stage cHL (Stage IIB, III and IV)
Number analyzed (Participants) | 51
Percent of Participants | 66.7 [52.1 to 79.2]

22. Post Hoc Outcome: Objective Response Rate (ORR) Based on IRRC Assessments in Cohorts A, B, and C Extended Collection
Description: Represents an updated version of the primary endpoint to include additional data collection that occurred after the primary completion date. (Assessments were made until 30 Nov 2022). Clinical benefit of nivolumab, as measured by ORR per IRRC assessment, and defined as percent of participants achieving either complete remission (CR) or partial remission (PR) according to the 2007 IWG criteria. For cohort A and B, if the bone marrow was involved by lymphoma before treatment, the infiltrate must have cleared on repeat bone marrow biopsy. For cohort C, no evidence of FDG-avid disease in bone marrow was required in all patients in lieu of bone marrow aspirate/ biopsy. CR is the percent of participants with a best overall response (BOR) of CR (disappearance of all evidence of disease) according to the 2007 IWG criteria. PR is the percent of participants with a best overall response (BOR) of PR (regression of measurable disease and no new sites) according to the 2007 IWG criteria.
Time Frame: From first dose to the date of initial objectively documented progression or the date of subsequent therapy, whichever occurred first (up to approximately 100 months)
Population: All treated Cohort A, B and C participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Post-Transplant, Never Taken Brentuximab Vedotin | Cohort B: Post Transplant, Brentuximab Vedotin Taken Post-Autologous Stem Cell Transplant | Cohort C: Post Transplant, Brentuximab Vedotin Taken Pre-and/or Post-Autologous Stem Cell Transplant
Number analyzed (Participants) | 63 | 80 | 100
Percentage of Participants | 65.1 [52.0 to 76.7] | 71.3 [60.0 to 80.8] | 75.0 [65.3 to 83.1]

ADVERSE EVENTS:
Time Frame: Participants were assessed for All-Cause Mortality from first dose until study completion (assessed up to approximately 100 months). SAEs and Other AEs were assessed from first dose to 100 days after last dose of study therapy (assessed for an average of 32 months up to maximum of 98 months).
Description: All-Cause Mortality and Serious and Other (Not Including Serious) Adverse Events is represented per dosage, per arm for Cohorts A, B, and C. This is to account for these events after the dosage and administration changes for nivolumab were implemented per revised protocol version 04c (dated 22-Aug-2019).
  Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
Groups:
- Cohort A: Post-Transplant, Never Taken Brentuximab Vedotin- Nivolumab 3 mg/kg; Cohort A: Post-Transplant, Never Taken Brentuximab Vedotin-Nivolumab 240 mg; Cohort A: Post-Transplant, Never Taken Brentuximab Vedotin-Nivolumab 480 mg; Cohort B: Post Transplant, Brentuximab Vedotin Taken Post-Stem Cell Transplant-Nivolumab 3 mg/kg; Cohort B: Post Transplant, Brentuximab Vedotin Taken Post-Stem Cell Transplant-Nivolumab 240 mg; Cohort B: Post Transplant, Brentuximab Vedotin Taken Post-Stem Cell Transplant- Nivolumab 480 mg; Cohort C: Post Transplant, Brentuximab Vedotin Pre-and/or Post-SC Transplant - Nivolumab 3 mg/kg; Cohort C: Post Transplant, Brentuximab Vedotin Pre-and/Post-Stem Cell Transplant - Nivolumab 240 mg; Cohort C: Post Transplant, Brentuximab Vedotin Pre-and/Post-Stem Cell Transplant - Nivolumab 480 mg: Nivolumab was administered at 3 mg/kg IV over 60 minutes on the first day of each 2-week cycle. Upon the implementation of revised protocol version 04c (dated 22-Aug-2019), participants were switched from a body weight-based dose of 3 mg/kg every 2 weeks to a flat dose of 480 mg every 4 weeks or a flat dose of 240 mg every 2 weeks. Nivolumab treatment was continued until unacceptable toxicity or disease progression.
Arm/Group | Cohort A: Post-Transplant, Never Taken Brentuximab Vedotin- Nivolumab 3 mg/kg | Cohort A: Post-Transplant, Never Taken Brentuximab Vedotin-Nivolumab 240 mg | Cohort A: Post-Transplant, Never Taken Brentuximab Vedotin-Nivolumab 480 mg | Cohort B: Post Transplant, Brentuximab Vedotin Taken Post-Stem Cell Transplant-Nivolumab 3 mg/kg | Cohort B: Post Transplant, Brentuximab Vedotin Taken Post-Stem Cell Transplant-Nivolumab 240 mg | Cohort B: Post Transplant, Brentuximab Vedotin Taken Post-Stem Cell Transplant- Nivolumab 480 mg | Cohort C: Post Transplant, Brentuximab Vedotin Pre-and/or Post-SC Transplant - Nivolumab 3 mg/kg | Cohort C: Post Transplant, Brentuximab Vedotin Pre-and/Post-Stem Cell Transplant - Nivolumab 240 mg | Cohort C: Post Transplant, Brentuximab Vedotin Pre-and/Post-Stem Cell Transplant - Nivolumab 480 mg | Cohort D: Newly Diagnosed, Previously Untreated Advanced Stage cHL (Stage IIB, III and IV)
All-Cause Mortality (participants affected / at risk) | 14/46 | 3/9 | 0/8 | 25/75 | 0/3 | 0/2 | 31/84 | 4/13 | 0/3 | 5/51
Serious Adverse Events (participants affected / at risk) | 10/46 | 3/9 | 1/8 | 30/75 | 0/3 | 1/2 | 33/84 | 8/13 | 3/3 | 12/51
Other Adverse Events (participants affected / at risk) | 46/46 | 9/9 | 8/8 | 75/75 | 3/3 | 2/2 | 80/84 | 13/13 | 3/3 | 50/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Post-Transplant, Never Taken Brentuximab Vedotin- Nivolumab 3 mg/kg (N=46) | Cohort A: Post-Transplant, Never Taken Brentuximab Vedotin-Nivolumab 240 mg (N=9) | Cohort A: Post-Transplant, Never Taken Brentuximab Vedotin-Nivolumab 480 mg (N=8) | Cohort B: Post Transplant, Brentuximab Vedotin Taken Post-Stem Cell Transplant-Nivolumab 3 mg/kg (N=75) | Cohort B: Post Transplant, Brentuximab Vedotin Taken Post-Stem Cell Transplant-Nivolumab 240 mg (N=3) | Cohort B: Post Transplant, Brentuximab Vedotin Taken Post-Stem Cell Transplant- Nivolumab 480 mg (N=2) | Cohort C: Post Transplant, Brentuximab Vedotin Pre-and/or Post-SC Transplant - Nivolumab 3 mg/kg (N=84) | Cohort C: Post Transplant, Brentuximab Vedotin Pre-and/Post-Stem Cell Transplant - Nivolumab 240 mg (N=13) | Cohort C: Post Transplant, Brentuximab Vedotin Pre-and/Post-Stem Cell Transplant - Nivolumab 480 mg (N=3) | Cohort D: Newly Diagnosed, Previously Untreated Advanced Stage cHL (Stage IIB, III and IV) (N=51)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 3 | 0 | 1 | 3 | 0 | 0 | 3
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute graft versus host disease (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Graft versus host disease (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Device related sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Febrile infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatitis A (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lyme disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Meningitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 5 | 0 | 0 | 5 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respirovirus test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Follicular lymphoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 2 | 0 | 0 | 4 | 0 | 0 | 0
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral T-cell lymphoma unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Post-Transplant, Never Taken Brentuximab Vedotin- Nivolumab 3 mg/kg (N=46) | Cohort A: Post-Transplant, Never Taken Brentuximab Vedotin-Nivolumab 240 mg (N=9) | Cohort A: Post-Transplant, Never Taken Brentuximab Vedotin-Nivolumab 480 mg (N=8) | Cohort B: Post Transplant, Brentuximab Vedotin Taken Post-Stem Cell Transplant-Nivolumab 3 mg/kg (N=75) | Cohort B: Post Transplant, Brentuximab Vedotin Taken Post-Stem Cell Transplant-Nivolumab 240 mg (N=3) | Cohort B: Post Transplant, Brentuximab Vedotin Taken Post-Stem Cell Transplant- Nivolumab 480 mg (N=2) | Cohort C: Post Transplant, Brentuximab Vedotin Pre-and/or Post-SC Transplant - Nivolumab 3 mg/kg (N=84) | Cohort C: Post Transplant, Brentuximab Vedotin Pre-and/Post-Stem Cell Transplant - Nivolumab 240 mg (N=13) | Cohort C: Post Transplant, Brentuximab Vedotin Pre-and/Post-Stem Cell Transplant - Nivolumab 480 mg (N=3) | Cohort D: Newly Diagnosed, Previously Untreated Advanced Stage cHL (Stage IIB, III and IV) (N=51)
Anaemia (Blood and lymphatic system disorders) | 4 | 1 | 1 | 12 | 0 | 0 | 18 | 2 | 0 | 9
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 4 | 1 | 0 | 7 | 0 | 0 | 9 | 2 | 0 | 28
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 3 | 0 | 0 | 14 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 3 | 0 | 1 | 1 | 1 | 0 | 3 | 1 | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 7 | 0 | 0 | 1 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 1 | 4 | 0 | 0 | 1 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 3 | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 3
Hypothyroidism (Endocrine disorders) | 7 | 1 | 1 | 9 | 0 | 0 | 7 | 2 | 0 | 8
Primary hypothyroidism (Endocrine disorders) | 1 | 0 | 1 | 3 | 0 | 0 | 1 | 1 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 3 | 1 | 0 | 7 | 0 | 0 | 1
Eye disorder (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Mydriasis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Swelling of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Vision blurred (Eye disorders) | 3 | 1 | 0 | 1 | 0 | 0 | 4 | 0 | 1 | 4
Visual field defect (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 7 | 1 | 0 | 14 | 2 | 1 | 13 | 0 | 0 | 4
Abdominal pain upper (Gastrointestinal disorders) | 6 | 3 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 1
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 7 | 2 | 1 | 14 | 1 | 1 | 15 | 0 | 1 | 18
Diarrhoea (Gastrointestinal disorders) | 26 | 3 | 5 | 37 | 1 | 2 | 25 | 6 | 1 | 17
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 0 | 3 | 0 | 0 | 4 | 1 | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 4 | 0 | 1 | 5 | 0 | 0 | 5 | 0 | 1 | 4
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 5 | 0 | 0 | 1 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 3 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 7 | 0 | 0 | 4 | 0 | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3
Nausea (Gastrointestinal disorders) | 14 | 1 | 5 | 20 | 1 | 1 | 19 | 1 | 1 | 31
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Steatorrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 5 | 0 | 1 | 3 | 0 | 0 | 4 | 0 | 0 | 12
Toothache (Gastrointestinal disorders) | 2 | 1 | 1 | 5 | 0 | 0 | 2 | 0 | 1 | 3
Vomiting (Gastrointestinal disorders) | 11 | 2 | 5 | 18 | 0 | 1 | 19 | 1 | 1 | 15
Asthenia (General disorders) | 4 | 1 | 2 | 9 | 0 | 0 | 3 | 1 | 0 | 7
Chest discomfort (General disorders) | 2 | 1 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 2
Chest pain (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 4
Chills (General disorders) | 2 | 3 | 1 | 4 | 0 | 0 | 4 | 3 | 0 | 6
Fatigue (General disorders) | 19 | 5 | 3 | 36 | 1 | 2 | 27 | 2 | 2 | 19
Feeling cold (General disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Influenza like illness (General disorders) | 2 | 0 | 3 | 5 | 2 | 1 | 2 | 1 | 2 | 0
Malaise (General disorders) | 1 | 2 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 1
Mucosal dryness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 4 | 1 | 0 | 3 | 0 | 0 | 2 | 1 | 1 | 5
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 1
Oedema peripheral (General disorders) | 2 | 0 | 0 | 6 | 0 | 0 | 11 | 1 | 0 | 2
Pain (General disorders) | 2 | 0 | 0 | 6 | 0 | 0 | 4 | 0 | 0 | 3
Peripheral swelling (General disorders) | 1 | 0 | 2 | 4 | 1 | 0 | 3 | 0 | 0 | 0
Pyrexia (General disorders) | 12 | 5 | 3 | 33 | 1 | 2 | 29 | 2 | 1 | 20
Thirst (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Venoocclusive liver disease (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 2 | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 2
Seasonal allergy (Immune system disorders) | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aeromonas infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atypical mycobacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 2 | 2 | 3 | 6 | 0 | 1 | 2 | 1 | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 5 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 4 | 0 | 0 | 3 | 1 | 0 | 1
Cystitis (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 3 | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 0 | 1
Gastric infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 1 | 3 | 1 | 0 | 1 | 0 | 0 | 2
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 4 | 0 | 2 | 2 | 0 | 0 | 3 | 2 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Infected skin ulcer (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 2 | 3 | 0 | 5 | 0 | 0 | 5 | 1 | 0 | 1
Lip infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymph gland infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 10 | 5 | 6 | 21 | 3 | 1 | 10 | 3 | 2 | 6
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 3 | 0 | 0 | 3 | 1 | 2 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 3
Pharyngitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 1 | 1 | 13 | 2 | 1 | 6 | 1 | 1 | 3
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 4 | 0 | 0 | 1 | 1 | 0 | 3
Rhinitis (Infections and infestations) | 1 | 3 | 1 | 6 | 0 | 0 | 3 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 3 | 1 | 6 | 0 | 1 | 4 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 11 | 1 | 3 | 28 | 1 | 0 | 18 | 3 | 0 | 6
Urinary tract infection (Infections and infestations) | 3 | 0 | 1 | 7 | 0 | 0 | 3 | 1 | 1 | 1
Viral infection (Infections and infestations) | 1 | 0 | 0 | 5 | 2 | 0 | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 6 | 0 | 0 | 13 | 1 | 1 | 9 | 1 | 1 | 16
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 6 | 2 | 2 | 11 | 0 | 0 | 9 | 0 | 0 | 3
Amylase increased (Investigations) | 2 | 1 | 0 | 7 | 0 | 1 | 3 | 1 | 0 | 3
Aspartate aminotransferase increased (Investigations) | 4 | 1 | 2 | 9 | 0 | 0 | 10 | 0 | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 2 | 1 | 0 | 6 | 0 | 0 | 8 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 4 | 0 | 1 | 2 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 1 | 0 | 6 | 0 | 0 | 3 | 0 | 0 | 1
Blood thyroid stimulating hormone increased (Investigations) | 1 | 1 | 0 | 3 | 0 | 0 | 2 | 1 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Lipase increased (Investigations) | 4 | 1 | 1 | 16 | 0 | 1 | 4 | 1 | 1 | 2
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 2 | 0 | 0 | 3 | 0 | 0 | 5 | 0 | 0 | 3
Neutrophil count decreased (Investigations) | 0 | 0 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 10
Platelet count decreased (Investigations) | 5 | 0 | 0 | 1 | 1 | 0 | 3 | 2 | 0 | 1
SARS-CoV-2 test positive (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sputum abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 3 | 0 | 3 | 6 | 0 | 1 | 4 | 0 | 0 | 1
Weight increased (Investigations) | 3 | 1 | 1 | 7 | 0 | 1 | 8 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 3 | 0 | 1 | 3 | 0 | 0 | 3 | 0 | 0 | 9
Decreased appetite (Metabolism and nutrition disorders) | 5 | 3 | 2 | 11 | 0 | 1 | 7 | 0 | 0 | 3
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 8 | 0 | 0 | 7 | 0 | 0 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 6 | 0 | 0 | 4 | 0 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 5 | 0 | 0 | 4 | 1 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2 | 0 | 0 | 6 | 0 | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 4 | 2 | 27 | 1 | 1 | 15 | 1 | 1 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 1 | 2 | 17 | 1 | 1 | 12 | 0 | 0 | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 3 | 0 | 1 | 8
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 4 | 1 | 0 | 1 | 0 | 0 | 1
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 11 | 0 | 0 | 5 | 1 | 0 | 1
Muscle swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 2 | 0 | 0 | 4 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 1 | 2 | 11 | 1 | 1 | 9 | 0 | 0 | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 6 | 0 | 0 | 7 | 1 | 0 | 3
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Convulsions local (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 6 | 0 | 1 | 10 | 1 | 0 | 7 | 0 | 0 | 8
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 14 | 3 | 2 | 15 | 0 | 0 | 13 | 3 | 2 | 7
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 5 | 0 | 0 | 1 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 2 | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 0 | 3
Migraine (Nervous system disorders) | 1 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Migraine with aura (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 3 | 1 | 0 | 9 | 0 | 1 | 3 | 1 | 0 | 5
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 3 | 0 | 1 | 2 | 0 | 0 | 4
Polyneuropathy (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 3 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1
Tremor (Nervous system disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 5 | 0 | 1 | 5 | 0 | 1 | 3
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 2 | 0 | 0 | 5 | 0 | 1 | 4 | 0 | 1 | 1
Generalised anxiety disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 4 | 1 | 1 | 12 | 0 | 2 | 7 | 0 | 0 | 5
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 2 | 0 | 0 | 4 | 0 | 0 | 3 | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Menopausal symptoms (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 5 | 4 | 31 | 0 | 1 | 28 | 5 | 2 | 13
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 1 | 0 | 0 | 2 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1 | 14 | 0 | 1 | 13 | 3 | 0 | 6
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 3 | 0 | 0 | 3 | 1 | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 1 | 0 | 0
Increased viscosity of upper respiratory secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9 | 0 | 5 | 9 | 0 | 1 | 8 | 1 | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 2 | 14 | 1 | 1 | 11 | 1 | 0 | 2
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paranasal sinus inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 6 | 0 | 0 | 4 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 3 | 6 | 0 | 1 | 4 | 1 | 0 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 4 | 0 | 0 | 4 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 5 | 0 | 0 | 8 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3 | 3 | 0 | 0 | 4 | 0 | 0 | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 4 | 0 | 0 | 2 | 0 | 0 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 3 | 0 | 0 | 2 | 1 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0 | 4 | 6 | 0 | 0 | 5 | 0 | 1 | 4
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 1 | 1 | 1 | 0 | 1 | 4 | 3 | 0 | 3
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 3 | 1 | 4 | 0 | 0 | 4 | 0 | 0 | 1
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 3 | 1 | 22 | 1 | 1 | 14 | 3 | 1 | 12
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 12 | 0 | 2 | 21 | 1 | 0 | 13 | 2 | 1 | 13
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 0 | 0 | 4 | 1 | 1 | 1 | 0 | 0 | 3
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 3 | 0 | 0 | 3 | 0 | 0 | 1
Flushing (Vascular disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 4 | 1 | 1 | 1
Hypertension (Vascular disorders) | 2 | 0 | 0 | 5 | 1 | 0 | 2 | 0 | 0 | 2
Lymphoedema (Vascular disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral venous disease (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Superficial vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication

DOCUMENTS (2):
  • Study Protocol (2019-08-22): https://cdn.clinicaltrials.gov/large-docs/38/NCT02181738/Prot_002.pdf
  • Statistical Analysis Plan (2018-06-08): https://cdn.clinicaltrials.gov/large-docs/38/NCT02181738/SAP_001.pdf